CLINICAL TRIAL: NCT00514046
Title: Phase I/II Trial of Vandetanib (ZD6474, ZACTIMA) in Children and Adolescents With Hereditary Medullary Thyroid Carcinoma
Brief Title: Vandetanib to Treat Children and Adolescents With Medullary Thyroid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brigitte Widemann, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070189; 07-C-0189
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Medullary Thyroid Carcinoma; Multiple Endocrine Neoplasia Type 2A; Multiple Endocrine Neoplasia Type 2B
Keywords: Multiple Endocrine Neoplasia; Medullary Thyroid Carcinoma; Molecularly-Targeted Therapy; Pediatric; Pharmacokinetics
MeSH Terms: conditions — Carcinoma, Medullary; Multiple Endocrine Neoplasia Type 2a; Multiple Endocrine Neoplasia Type 2b; Multiple Endocrine Neoplasia | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vandetanib (Experimental): Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 150 mg/m^2/day.
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — once daily continuously (28 day cycles)
  Other Names: Caprelsa

SUMMARY:
Background:

* Medullary thyroid carcinoma (MTC) is common in people with a genetic disorder called multiple endocrine neoplasia (MEN).
* Vandetanib is an experimental drug that blocks a defective protein receptor (rearranged during transfection (RET) receptor) found on the surface of cancer cells in people with MEN. It is thought that this protein is a primary cause of MTC in people with MEN.

Objectives:

* To study the activity of Vandetanib in children and adolescents with MEN-related MTC by measuring the change in tumor size, in blood levels of proteins produced the tumor (calcitonin and carcinoembryonic antigen (CEA) and in tumor-related diarrhea.
* To determine the safety and tolerability of Vandetanib in children and adolescents.
* To study how the body handles Vandetanib in children and adolescents.
* To determine the effect of Vandetanib on the survival of children and adolescents with MTC.

Eligibility:

-Children and adolescents 5 to 18 years of age with MTC whose tumor cannot be surgically removed or has grown back after treatment or has metastasized (spread beyond the thyroid gland).

Design:

* Patients take Vandetanib once a day in 28-day cycles. The first patients enrolled in the study are started on a low dose of Vandetanib to determine tolerability.
* Patients have periodic blood tests, electrocardiograms, and blood pressure measurements to look for side effects of Vandetanib.
* Blood tests and imaging scans (magnetic resonance imaging (MRI), computed tomography (CT), bone and octreoscan) are done every 8 weeks for the first 32 weeks of treatment and then every 16 weeks for the duration of the treatment period.
* Patients who have tumor-related diarrhea keep a daily record of the number and consistency of bowel movements.

DETAILED DESCRIPTION:
BACKGROUND:

Hereditary medullary thyroid carcinoma (MTC), which is a rare calcitonin-producing tumor arising from the parafollicular C cells of the thyroid, is often a manifestation of multiple endocrine neoplasia (MEN) types 2A and 2B and can be detected in children as young as five years in MEN 2A and one year in those with MEN 2B

MEN results from an activating mutation in the rearranged during transfection (RET) proto-oncogene resulting in a constitutively activated receptor tyrosine kinase (RTK)

Vandetanib is an orally bioavailable multi-RTK inhibitor that blocks the mutant RET gene product and has anti-tumor activity in adults with hereditary MTC

OBJECTIVES:

To assess the activity of vandetanib in children and adolescents with hereditary MTC using Response Evaluation Criteria in Solid Tumors (RECIST) (primary endpoint), tumor biomarkers and tumor-related diarrhea

To assess the safety and tolerance of vandetanib in children and adolescents at a dose equivalent to the recommended dose in adults

To assess the pharmacokinetics of vandetanib at steady state in children and adolescents

Secondary objectives include monitoring progression-free and overall survival, assessing RET, epidermal growth factor receptor (EGFR), Vascular endothelial growth factor (VEGFR) and somatostatin receptor expression in archival tumor tissue, assessing changes in deoxyribonucleic acid (DNA) mutations in RET in tumor tissue vs germ line in PBMC and after treatment; assessing gene expression and gains/losses of DNA in tumor tissue at baseline, during treatment and at the time of progression; establishment of pediatric MTC cell lines sensitive and resistant cells lines in vitro

ELIGIBILITY:

Children and adolescents 5 to 18 years of age (inclusive) with unresectable, recurrent or metastatic hereditary medullary thyroid carcinoma

Measurable disease by RECIST (Response Evaluation Criteria in Solid Tumors)

DESIGN:

Vandetanib will be administered as a once daily dose, continuously (1 cycle equals 28 days) at a dose of 150 mg,m(2), per day

To ensure the safety of the adult dose in children and adolescents, a limited intra-patient dose escalation will be performed in the initial cohort of patients, with older patients (13 to18 yrs) being studied before younger patients (5 to12 yrs)

Patients wil be enrolled at a dose of 100mg, m(2), per day (180 mg per day in adults) for two 28 day cycles and escalated to 150 mg, m(2), per day (270 mg, per day in adults) on cycle 3, if dose limiting toxicity was not observed at the lower dose. If the 150mg, m(2), per day dose level is tolerable on cycles 3 and 4, all subsequent patients will be enrolled at this dose level

Pharmacokinetics of vandetanib will be studied at steady state at the end of cycle 2 and trough levels will be obtained prior to the second dose on cycle 1, and on day 1 of cycles 2-5.

Responsible of measurable tumors will be assessed by RECIST. Biomarker and clinical response will also be monitored. Twenty one patients will be studied to determine if the response rate in children and adolescents with hereditary MTC is consistent with the 28 percent objective response rate in adults

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Participants must be 5 to 18 years of age, inclusive. The first cohort of 3 to 6 participants enrolled on the trial will be at least 13 years of age.

Diagnosis: Hereditary (Multiple endocrine neoplasia, type 2A (MEN 2A) or Multiple endocrine neoplasia, type 2B (MEN 2B) medullary thyroid carcinoma (histologically confirmed) that is unresectable, recurrent or metastatic. Participants must have previously had a characteristic germline mutation in the rearranged during transfection (RET) proto-oncogene documented. Results of the germline mutation testing will be obtained from the referring institution.

Participants must have measurable disease as defined in Response Evaluation Criteria in Solid Tumors (RECIST) as the presence of at least one lesion that can be accurately measured in at least one dimension with longest diameter of at least 20 mm using conventional techniques or at least 10 mm with spiral computed tomography (CT) scan. Superficial (easily palpable) lymph nodes will be considered measurable.

Participants must be able to take one of the oral formulations of vandetanib.

Prior therapy: There are no standard chemotherapy regimens known to be effective for medullary thyroid carcinoma (MTC). Therefore, previously untreated participants are eligible if their tumor(s) are not surgically resectable.

Participants must be at least 4 weeks from prior surgical procedures and surgical incisions must be healed.

Participants must have had their last fraction of external beam radiation therapy at least 4 weeks prior to enrollment.

Participants must have had their last dose of cytotoxic chemotherapy at least 28 days prior to enrollment, their last dose of biological therapy, such as biological response modifiers (e.g., cytokines), immunomodulatory agents, vaccines, differentiating agents, used to treat their cancer at least 7 days prior to enrollment, their last dose of a monoclonal antibody at least 30 days prior to enrollment, and their last dose of any investigational agent at least 30 days prior to enrollment.

Participants must have received their last dose of short acting colony stimulating factor, such as filgrastim or sargramostim at least 72 hours prior to enrollment and their last dose of long-acting colony stimulating factors, such as polyethylene glycol (PEG)-filgrastim at least 7 days prior to enrollment.

Participants must have recovered from the acute toxic effects of prior therapy to a grade 1 (Common Terminology Criteria for Adverse Events (CTCAE) v.3.0) level prior to enrollment.

Performance Status: Lansky (for participants 10 years of age or younger) or Karnofsky (for participants older than 10 years) performance score greater than 50

Concomitant Medications:

Participants who have previously had a thyroidectomy should be on thyroid hormone replacement therapy.

Hematological Function: The peripheral absolute neutrophil count must be at least 1,500 micro liters and the platelet count must be at least 100,000 micro liters within 72 hours prior to enrollment.

Coagulation: Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) must not be more than 1.5 x ULN within 72 hours prior to enrollment. PT and PTT should drawn by venipuncture, rather than from a central venous catheter when feasible.

Hepatic Function:

Bilirubin must not be more than 1.5 x ULN and the aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must not be more than 2.5 x ULN within 72 hours prior to enrollment. AST and ALT may be up to 5 x ULN within 72 hours prior to enrollment in participants with hepatic metastases.

Renal Function: Participants must have an age-adjusted normal serum creatinine or a creatinine clearance of at least 60 ml/min/1.73 m^2.

Birth Control: Participants of child-bearing or child-fathering potential must be willing to use a medically effective form of birth control, which includes abstinence, while taking vandetanib and for 2 months after the last dose.

Negative pregnancy test for women of childbearing potential.

Informed Consent: Participants who are 18 years of age or legal guardians of participants who are younger than 18 years must sign an informed consent for the Pediatric Oncology Branch (POB) Screening Protocol prior to participating in studies required to determine eligibility for this trial. After confirmation of eligibility, participants or legal guardians of minor participants must sign an informed consent document for this trial, indicating that they are aware of the investigational nature of the proposed treatment, the risks and benefits of participating and the alternatives to participating.

EXCLUSION CRITERIA:

Pregnant or breast feeding females because the anti-angiogenic properties of vandetanib may be harmful to the developing fetus or nursing infant.

Participants with pheochromocytoma as evidenced by elevated plasma free metanephrines.

Electrolytes: Participants with a serum potassium less than 3.5 mmol/L or a serum calcium or magnesium below the lower limits of normal. Correction of these electrolyte abnormalities with supplements is allowed.

Cardiac:

Participants with a history of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, uncontrolled atrial fibrillation, left bundle branch block) that is symptomatic or requires treatment (except for controlled atrial fibrillation)

Participants with a history of congenitally prolonged Corrected QT Interval (QTc), a first degree relative with unexplained sudden death under 40 years of age, or a measured QTc (Bazett's correction) longer than 480 msec on electrocardiogram (ECG). ECGs should be performed after correction of electrolyte abnormalities. Participants with a prolonged QTc should have a repeat ECG at least 24 hour after the first, and the mean of the 2 QTcs should not exceed 480 msec.

Participants who experienced QTc prolongation with other medications requiring discontinuation of that medication.

Participants receiving a medication that has a known risk of QTc prolongation within 14 days (28 days for levomethadyl) of enrollment.

Hypertension: Diastolic blood pressure above the 95% for age on at least 2 of 3 measurements with an appropriate-size cuff or patients who are currently taking anti-hypertensive therapy.

Other clinically severe or uncontrolled systemic illness that could compromise the participants ability to tolerate vandetanib or could compromise study procedures or endpoints.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07-20 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We wish to share IPD via two citations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Indefinitely.

REFERENCES:
- [Background] Holden SN, Eckhardt SG, Basser R, de Boer R, Rischin D, Green M, Rosenthal MA, Wheeler C, Barge A, Hurwitz HI. Clinical evaluation of ZD6474, an orally active inhibitor of VEGF and EGF receptor signaling, in patients with solid, malignant tumors. Ann Oncol. 2005 Aug;16(8):1391-7. doi: 10.1093/annonc/mdi247. Epub 2005 May 19. PMID 15905307
- [Background] Marsh DJ, Learoyd DL, Robinson BG. Medullary thyroid carcinoma: recent advances and management update. Thyroid. 1995 Oct;5(5):407-24. doi: 10.1089/thy.1995.5.407. PMID 8563482
- [Result] Fox E, Widemann BC, Chuk MK, Marcus L, Aikin A, Whitcomb PO, Merino MJ, Lodish M, Dombi E, Steinberg SM, Wells SA, Balis FM. Vandetanib in children and adolescents with multiple endocrine neoplasia type 2B associated medullary thyroid carcinoma. Clin Cancer Res. 2013 Aug 1;19(15):4239-48. doi: 10.1158/1078-0432.CCR-13-0071. Epub 2013 Jun 13. PMID 23766359
- [Result] Kraft IL, Akshintala S, Zhu Y, Lei H, Derse-Anthony C, Dombi E, Steinberg SM, Lodish M, Waguespack SG, Kapustina O, Fox E, Balis FM, Merino MJ, Meltzer PS, Glod JW, Shern JF, Widemann BC. Outcomes of Children and Adolescents with Advanced Hereditary Medullary Thyroid Carcinoma Treated with Vandetanib. Clin Cancer Res. 2018 Feb 15;24(4):753-765. doi: 10.1158/1078-0432.CCR-17-2101. Epub 2017 Nov 29. PMID 29187393
- [Result] Allen, T., Bedoya, S.Z., Glod, J., Widemann, B., Wiener, L. Baseline Characteristics of Adolescents and Young Adults with Medullary Thyroid Cancer and MEN-2B: Data from the Rare Tumor Initiative at the National Cancer Institute. International Psycho-Oncology Society's 21st World Congress, Banff, Canada, September, 2019, Journal of Psychosocial Oncology Research and Practice, 1(1): 5.
- [Derived] Lodish M, Gkourogianni A, Bornstein E, Sinaii N, Fox E, Chuk M, Marcus L, Akshintala S, Balis F, Widemann B, Stratakis CA. Patterns of thyroid hormone levels in pediatric medullary thyroid carcinoma patients on vandetanib therapy. Int J Pediatr Endocrinol. 2015;2015(1):3. doi: 10.1186/1687-9856-2015-3. Epub 2015 Feb 16. PMID 25972901
- [Derived] Nella AA, Lodish MB, Fox E, Balis FM, Quezado MM, Whitcomb PO, Derdak J, Kebebew E, Widemann BC, Stratakis CA. Vandetanib successfully controls medullary thyroid cancer-related Cushing syndrome in an adolescent patient. J Clin Endocrinol Metab. 2014 Sep;99(9):3055-9. doi: 10.1210/jc.2013-4340. Epub 2014 Mar 11. PMID 24617713
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0189.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Vandetanib: First 100 mg/m^2, Then 150 mg/m^2: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 150 mg/m^2.
- Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 150 mg/m^2, followed by 67 mg/m^2.
- Vandetanib 100 mg/m^2: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day.
- Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 150 mg/m^2, followed by 100 mg/m^2.
- Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 63 mg/m^2, then 42 mg/m^2, then 21 mg/m^2, then 42 mg/m^2, followed by 21 mg/m^2.
- Vandetanib: First 100 mg/m^2, Then 70 mg/m^2: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 70 mg/m^2.
- Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 150 mg/m^2, followed by 200 mg/m^2.
- Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 100 mg/m^2/day, then 150 mg/m^2, then 100 mg/m^2, then 150 mg/m^2, then 100 mg/m^2, followed by 150 mg/m^2.
- Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg: All participants who received a starting dose of Vandetanib administered as a once daily dose, continuously (1 cycle = 28 days) at a dose of 150 mg/m^2/day, then 100 mg/m^2.
Period: Overall Study
Arm/Group | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg | Vandetanib 100 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg
Started | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not Completed | 3 | 1 | 5 | 0 | 1 | 1 | 0 | 1 | 1
Not completed — transferred to another protocol | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Getting vandetanib via the REMS program | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Disease progression on study | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg | Vandetanib 100 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg | Total
Number analyzed (Participants) | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 17
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.14 (2.07) | 15.4 (0) | 12.52 (2.81) | 16.7 (0) | 12.1 (0) | 17.3 (0) | 13.2 (0) | 11.3 (0) | 16.8 (0) | 14.50 (2.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 9
  Male | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 3 | 1 | 4 | 0 | 1 | 1 | 1 | 0 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 5 | 1 | 4 | 1 | 1 | 1 | 1 | 1 | 0 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Baseline Performance Status [Median (Full Range); unit: scores on a scale] — Karnofsky criteria for patients >10 year: 100 is normal, no complaints, no evidence of disease; 90 is able to carry on normal activity, minor signs or symptoms of disease; and 80 is normal activity with effort, some signs or symptoms of disease. Lansky criteria for children ≤10 years: 100 is fully active, normal; 90 is minor restrictions in physically strenuous activity; and 80 is active, but tires more quickly.
  scores on a scale | 100 [90 to 100] | 80 [80 to 80] | 80 [80 to 100] | 80 [80 to 80] | 100 [100 to 100] | 90 [90 to 90] | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100] | 100 [80 to 100]
Calcitonin (CTN) at Enrollment [Number; unit: pg/mL] — Calcitonin upper limit of normal is <10 pg/mL. A ≥50% increase in CTN from baseline indicates tumor growth or progression.
  pg/mL
    Patient 1 | 0 | 18,300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 2 | 67,100 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 3 | 0 | 0 | 4,500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 4 | 0 | 0 | 25,900 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 5 | 0 | 0 | 18,900 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 6 | 0 | 0 | 0 | 4,600 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 7 | 0 | 0 | 0 | 0 | 0 | 2,000 | 0 | 0 | 0 | 0
    Patient 8 | 0 | 0 | 0 | 0 | 3,500 | 0 | 0 | 0 | 0 | 0
    Patient 9 | 500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 10 | 0 | 0 | 57,800 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 11 | 0 | 0 | 0 | 0 | 0 | 0 | 13,300 | 0 | 0 | 0
    Patient 12 | 6,900 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 13 | 24,200 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 14 | 21,400 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 800 | 0 | 0
    Patient 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47.700 | 0
    Patient 17 | 0 | 0 | 16,064 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carcinoembryonic Antigen (CEA) at Enrollment [Number; unit: ng/mL] — CEA upper limit of normal is 4.6 ng/mL. A ≥50% increase in CEA from baseline indicates tumor growth or progression.
  ng/mL
    Patient 1 | 0 | 341.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 2 | 130.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 3 | 0 | 0 | 444.2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 4 | 0 | 0 | 247.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 5 | 0 | 0 | 60.2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 6 | 0 | 0 | 0 | 17.7 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 7 | 0 | 0 | 0 | 0 | 0 | 6.8 | 0 | 0 | 0 | 0
    Patient 8 | 0 | 0 | 0 | 0 | 115.5 | 0 | 0 | 0 | 0 | 0
    Patient 9 | 8.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 10 | 0 | 0 | 801.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 11 | 0 | 0 | 0 | 0 | 0 | 0 | 133.4 | 0 | 0 | 0
    Patient 12 | 28.4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 13 | 244.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 14 | 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Patient 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5.1 | 0 | 0
    Patient 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 60 | 0
    Patient 17 | 0 | 0 | 863 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is the highest dose of Vandetanib tolerated at which a participant experienced a dose limiting toxicity (DLT) during the first two cycles of drug.
Time Frame: During Cycle 1 and Cycle 2, approximately 56 days
Measure: Number; unit: mg/m^2/day
Groups:
- All Participants: All participants who received Vandetanib 100mg/m^2 and 150mg/m^2.
Arm/Group | All Participants
Number analyzed (Participants) | 17
mg/m^2/day | 100

2. Primary Outcome: Overall Percentage of Participants With an Objective Response Defined as a Complete Response (CR) or Partial Response (PR)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Progressive Disease is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Patients were evaluated for response after every 2 cycles x 4 (prior to cycles 1, 3, 5, 7, and 9) and then after every 4 cycles X 1 (prior to cycle 13) and then every 6 cycles (prior to cycle 19, 25, 31, etc). Response was followed for an median of 59 mon
Population: This is the analysis of all 17 patients across dosing groups. Because dosing for each patient was adjusted over time based on toxicity and often patients did not have a radiographic response until they had a number of cycles of treatment, we combined all dosing groups when calculating response rate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 17
percentage of participants | 59 [33 to 82]

3. Secondary Outcome: Number of Participants With an Increase or Decrease in Carcinoembryonic Antigen (CEA) Biomarker Response
Description: Blood was collected from participants and measured with an Axsym Analyzer then Immulite CEA method and assessed by the following response criteria. Partial Response (PR) is a ≥50% decrease in the CEA level relative to the baseline level, confirmed with a repeat CEA level at least 4 weeks apart. Progression (P) is a ≥50% increase in the CEA relative to the prior value on 2 consecutive measurements at least 4 weeks apart. The patient must have been taking vandetanib for 4 weeks prior to the first measurements and must have continued to take the drug through the time that the second measurement was drawn. Stable (S) is a <50% increase or decrease in CEA level relative to the baseline level.
Time Frame: Every 2 cycles x 4 (prior to cycles 1, 3, 5, 7 and 9), prior to cycle 13, and then every 6 cycles (prior to cycle 19, 25, 31, etc). Patients were followed for response for a median of 59 months.
Population: Patients with CEA <2x upper limit of normal at baseline were not evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg | Vandetanib 100 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg
Number analyzed (Participants) | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1
Participants
  <50% decrease/<50% increase | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  >50% increase | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ≥50% decrease | 3 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 1
  Not Evaluable (NE) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

4. Secondary Outcome: Percent Change in Calcitonin (CTN) Biomarker Response After Cycle 1
Description: Blood was collected from participants and measured with an Chemiluminescence immunoassay. Calcitonin upper limit of normal is <10 pg/mL. A decline in CTN is defined as a ≥50% increase (e.g. tumor growth or progression) in the CTN level after treatment in cycle 1.
Time Frame: Cycle 1 (28 days)
Population: This data was only analyzed after cycle 1 and was not collected from the patient who received 150mg/m^2 dosing during cycle 1. All other patients received 100mg/m^2 dosing during cycle 1.
Measure: Number (95% Confidence Interval); unit: percent change in calcitonin
Groups:
- All Participants: All participants who received Vandetanib 100mg/m^2 during the first cycle.
Arm/Group | All Participants
Number analyzed (Participants) | 16
percent change in calcitonin | -59 [-84 to -34]

5. Secondary Outcome: Area Under the Concentration Time Curve (AUC 0-24h)
Description: The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: Cycle 1, Pre-dose and then 1, 2, 4, 6, 8, 10 and 24 hour post dose.
Population: All 11 subjects who had PK analysis were receiving a dose of 100mg/m^2/dose at the time that the PK analysis was done. All participants are grouped together because this data was performed during cycle 1 and was not collected for the patient who received 150mg/m^2 during cycle 1.
Measure: Median (Full Range); unit: mcg*h/mL
Arm/Group | All Participants
Number analyzed (Participants) | 11
mcg*h/mL | 16 [13.5 to 23.3]

6. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 142 months and 8 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg | Vandetanib 100 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg
Number analyzed (Participants) | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1
Participants | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1

7. Other Pre Specified Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: Hematologic Dose-Limiting Toxicity (H-DLT) is: Neutrophil count below 1,000/μL (grade 3) on 2 consecutive measurements drawn at least 72 hours apart OR a single neutrophil count below 500/μL (grade 4); Platelet count below 50,000/μL (grade 3) on 2 consecutive measurements drawn at least 72 hours apart OR a single platelet count below 25,000/μL (grade 4); A platelet transfusion administered when platelet count is below 50,000/μL is dose limiting thrombocytopenia, unless the transfusion is being administered for perioperative coverage; Grade 3 or 4 decrease in hemoglobin that can be corrected to at least 8.0 g/dl (grade 2) by transfusion of red blood cells is not a dose-limiting toxicity. Grade 3 or 4 hemolysis is a dose-limiting toxicity if it is judged to be vandetanib-related. Non-Hematologic Dose-Limiting Toxicity is any grade 3 or higher non-hematologic toxicity, with some exceptions such as Grade 3 nausea that is controlled by symptomatic treatment with anti-emetics.
Time Frame: up to Cycle 3 (each Cycle is 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg | Vandetanib 100 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg
Number analyzed (Participants) | 5 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 1
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 142 months and 8 days.
Arm/Group | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg | Vandetanib 100 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1 | 0/5 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/1 | 1/5 | 1/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1 | 4/5 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 (N=5) | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg (N=1) | Vandetanib 100 mg/m^2 (N=5) | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg (N=1) | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 (N=1) | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 (N=1) | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg (N=1) | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg (N=1) | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg (N=1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Gastroenteritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction, GI::Gallbladder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Gallbladder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib: First 100 mg/m^2, Then 150 mg/m^2 (N=5) | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 67mg (N=1) | Vandetanib 100 mg/m^2 (N=5) | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 100mg (N=1) | Vandetanib:First 100mg/m^2, Then 63mg, 42, 21, 42, & 21mg/m^2 (N=1) | Vandetanib: First 100 mg/m^2, Then 70 mg/m^2 (N=1) | Vandetanib: First 100mg/m^2, Then 150mg/m^2, Followed by 200mg (N=1) | Vandetanib:First 100mg/m^2, Then 150mg, 100, 150, 100, 150mg (N=1) | Vandetanib: First 150mg/m^2, Then 100mg/m^2, Followed by 150mg (N=1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (30) | 0 (0) | 3 (17) | 1 (2) | 1 (2) | 1 (8) | 1 (3) | 1 (5) | 1 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (10) | 1 (1) | 3 (11) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 1 (2) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 3 (6) | 1 (7) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (7) | 1 (2) | 3 (13) | 1 (5) | 0 (0) | 1 (7) | 0 (0) | 1 (4) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy/Immunology (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Other (Specify, "Intermittent facial pruritus/erythema w/watery eyes/nasal congestion)
Anorexia (Gastrointestinal disorders) | 3 (3) | 1 (3) | 3 (8) | 1 (1) | 1 (3) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 3 (12) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood/Bone Marrow - Other (Specify, "Mild Fe deficiency") (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone: spine-scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (8) | 1 (2) | 3 (9) | 1 (1) | 1 (5) | 1 (22) | 0 (0) | 1 (4) | 1 (1)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac General - Other (Specify, "+ grade 3/6 systolic ejection murmur") (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac General - Other (Specify ystolic Heart murmur) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (8) | 1 (9) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constitutional Symptoms - Other (Specify, Fever not specified, ANC unknown) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (7) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental: periodontal disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify,"2 cm clavicle mass nonmobile/tender to touch") (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify,"Abrasion to ant. Lt flank") (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify ,"Clubbing nail beds fingers & toes") (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, "Foot blister") (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify,"J uvenile Plantar Dermatosis") (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, "Several abrasions to the lower extremities") (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, "Soft/mobile nodule consistent w/ a cyst") (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Bil. thumb-nail changes (splitting/color change)) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Dermatitis) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Dermatitis plantar) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Dyshidrotic eczema) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Erythema GT site) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Erythema on the right side of thrach) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Follcullitis-RT upper shoulder,forearm) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Folliclitis, bug bites) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Folliculitis:chest & abdomen) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Hand & Foot syndrome:water blisters) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify Ingrown toe nail) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify ,Intermittent Granuloma tissue) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Intermittent paronychia secondary to ingrown toe nails) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Intermittent seborrheic dermatitis) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Lump under chin) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, Rt great toe erythema) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (55) | 1 (65) | 4 (166) | 1 (45) | 1 (18) | 1 (5) | 1 (54) | 1 (32) | 0 (0)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (3) | 1 (1) | 1 (4) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine - Other (Specify, "Cold intolerance") (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Endocrine - Other (Specify, Elevated parathyroid) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid dysfunction (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (8) | 1 (7) | 3 (7) | 1 (4) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (4) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu-like syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, "Healing sore on oral mucosa") (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, "Slight increase in borborygmi") (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, Borborygmi) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, Borborygmi: hyperactive bowel sounds) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, Duodenitis) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, Gastroenteritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, upset stomach / no diarrhea) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 3 (6) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI::Anus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU::Kidney (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU::Uterus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Specify, Quaiac test (+) x2) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Other (Specify, "Hepatitis w/ cholestatic component Intermittent obstruction/infection)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 3 (6) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 1 (4)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Oral Thrush) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Paronychia Lt foot) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Pharyngitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify,Pt had a "cold") (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Pt treated for UTI based on + urinestix") (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Rt great toe paronychia) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Seborrheic dermatitis scalp) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Specify,Staph aureus skin infection follicular rash) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Specify, Staphilococcus aureus abcesses + for MRSA) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify ,Tinea Pedis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Tinea circinata left hand) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, URI) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, URI nasal congestion/clear nasal discharge) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, URI:nasal congestion) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Specify, Viral gastroenteritis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Viral illness Acute Gastroenteritis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, Warts Rt knee) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Specify, parochyia Lt great toe) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bone (osteomyelitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Joint (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lip/perioral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Liver (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nose (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Ungual (nails) (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infection with unknown ANC::Bronchus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Dental-tooth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Kidney (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Middle ear (otitis media) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Pharynx (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Skin (cellulites) (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Trachea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Ungual (nails) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Vagina (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint-function (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Investigations) | 3 (12) | 1 (14) | 1 (2) | 0 (0) | 1 (8) | 1 (11) | 0 (0) | 0 (0) | 0 (0)
Lymphatics - Other (Specify ,lymphyadenopathy: cervical) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 1 (5) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (4) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 4 (10) | 1 (1) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 1 (1)
Metabolic/Laboratory - Other (Specify, Hyperphosphate) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other (Specify, Hyperphosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other (Specify, Metanephephrine) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other (Specify,Parathyroid, elevated) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other (Specify, Vit D defiency) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood alteration::Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration::Anxiety (Psychiatric disorders) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration::Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Specify, "Leg length discrepancy") (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Specify, "Limited ROM Lt hip") (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Specify, "Trauma Rt hip") (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Specify, Leg cramps) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Specify, Pectus carinatum) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (14) | 4 (8) | 1 (7) | 1 (3) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Neurology - Other (Specify, Tingling/pins/needles sensation from hip down when Pt lies on Lt side) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (6) | 1 (10) | 0 (0) | 1 (5) | 1 (11) | 1 (10) | 1 (1) | 1 (2) | 1 (2)
Ocular surface disease (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual - Other (Specify, keratoconus) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual - Other (Specify, Occasional tearing of her eyes after reading a lot) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0)
Pain - Other (Specify ,"Body aches") (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, Pain in rash) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, Pain ingrown toenails) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, Shooting pain Left 4 & 5th toes) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, Throat/pharynx/larynx) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (4) | 1 (5) | 2 (5) | 1 (3) | 1 (7) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain::Buttock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::External ear (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 5 (34) | 1 (15) | 1 (2) | 1 (16) | 1 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (3) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pain::Kidney (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Lymph node (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Oral-gums (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Pain NOS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Stomach (Gastrointestinal disorders) | 3 (5) | 1 (4) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Throat/pharynx/larynx (Gastrointestinal disorders) | 2 (2) | 1 (6) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Vagina (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (5) | 1 (1) | 0 (0)
Platelets (Investigations) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (11) | 0 (0) | 0 (0) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 5 (37) | 1 (2) | 4 (26) | 1 (5) | 1 (4) | 1 (4) | 1 (5) | 1 (2) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 5 (35) | 1 (1) | 3 (16) | 1 (3) | 1 (2) | 1 (9) | 1 (7) | 1 (1) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, "Cold symptoms: congestion") (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, Bronchitis infection) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, Cysts) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, Nasal congestion/Clear nasal discharge") (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (10) | 1 (6) | 2 (9) | 1 (4) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5 (11) | 1 (7) | 4 (9) | 1 (2) | 1 (1) | 1 (1) | 1 (5) | 1 (2) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Specify,"Burning on urination: dysuria") (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual/Reproductive Function - Other (Specify, Menorrhagia) (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual/Reproductive Function - Other (Specify, prolonged menstruation) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (diaphoresis) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 3 (6) | 1 (4) | 3 (6) | 1 (2) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular - Other (Specify, Lt LE les c/w localized pigmented purpura (capillaritis)) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (17) | 1 (2) | 4 (29) | 1 (7) | 1 (11) | 1 (6) | 1 (1) | 1 (2) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Weight loss (General disorders) | 1 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT00514046/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT00514046/ICF_001.pdf